CLINICAL TRIAL: NCT05603728
Title: An Open Label, Multi-Center, Retrospective and Prospective Evaluation of Shoulder Arthroplasty Clinical and Radiographic Outcomes
Brief Title: Exactech Shoulder Post Market Clinical Follow-up Study
Status: Recruiting | Type: Observational
Sponsor: Exactech (Industry)
Responsible Party: Sponsor
Other Study IDs: CR09-005
Record Dates: First submitted 2022-10-25; First posted 2022-11-03 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Osteo Arthritis Shoulders; Osteonecrosis; Rotator Cuff Tears; Rotator Cuff Tear Arthropathy; Ankylosing Spondylitis; Post-traumatic Osteoarthritis; Rheumatoid Arthritis; Fracture; Infections
MeSH Terms: conditions — Osteonecrosis; Rotator Cuff Injuries; Rotator Cuff Tear Arthropathy; Spondylitis, Ankylosing; Arthritis, Rheumatoid; Fractures, Bone; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to collect and evaluate long-term clinical and radiographic outcomes data in order to better understand the safety and performance of the shoulder arthroplasty over time. This study will follow subjects long-term for a minimum of 10-years, without an early-term restriction on the amount of time they will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Patient is indicated for shoulder arthroplasty (or has previously undergone shoulder arthroplasty)
* Patient is skeletelly mature
* Patient is expected to survive at least 2 years beyond surgery
* Patient is willing to participate by complying with pre- and postoperative visit requirements
* Patient is willing and able to read and sign a study informed consent form

Exclusion Criteria:

* Osteomyelitis of the proximal humerus or scapula; if a systemic infection or a secondary remote infection is suspected or confirmed, implantation should be delayed until infection is resolved
* Inadequate or malformed bone that precludes adequate support or fixation of the prosthesis
* Medial humeral bone loss resulting in compromised humeral stem fixation
* Proximal humeral bone loss extending distal to the surgical neck where there is compromised humeral stem fixation
* Neuromuscular disorders that do not allow control of the joint
* Significant injury to the brachial plexus
* Non-functional deltoid muscles
* Patient's age, weight, or activity level would cause the surgeon to expect early failure of the system
* The patient is unwilling or unable to comply with the post-operative care instructions
* Alcohol, drug, or other subtance abuse
* Any disease state that could adversaly affect the function or longevity of the implant
* Patient is pregnant
* Patient is a prisoner
* Patient is contraindicated for the surgery
* Revision cases in which a stemmed humeral component was used (Stemless Shoulder System)
* Metal allergy or sensitivity to the implants materials (Stemless Shoulder System)
* Acute fracture of the proximal humerus and displacement of the tuberosities, displaced three or four part fractures of the proximal humerus (hemi-arthroplasty), or acture fracture of the proximal humerus with failure of the glenohumeral joint (total anatomic shoulder arthroplasty) (Stemless Shoulder System)
* Acute fracture of the proximal humerus in combination with degenerative diseases of the glenohumeral joint and a grossly deficient, irreparable rotator cuff resulting in superior migration of the humeral head (reverse total shoulder arthroplasty) (Stemless Shoulder System)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who meet eligibility criteria - Patients who consent to participate to return for follow-up visits out to 10 years or longer
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2007-07-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Constant | Through study completion, an average of 1 per year
  Constant Shoulder Score - 100 points scale about pain, Activities of daily living, Strength test, and Range of Motions questions about shoulder where 100 % corresponds to the highest pain
ASES | Through study completion, an average of 1 per year
  American Shoulder and Elbow Surgeons Score (ASES) - 100 points scale about shoulder pain and performance evaluation in activities of daily living where 100 indicates the best shoulder condition
Oxford Score (may be used as an optional form for surgeons in the United Kingdom) | Through study completion, an average of 1 per year
  Oxford Shoulder Score (OSS) - 12 questions assessing outcomes of shoulder surgery and its impact on patients' quality of life of degenerative conditions such as arthritis and rotator cuff problems - Maximum score is 60 and indicates greater degree of disability
TESS (may be used as specific forms related to the pre-operative condition/diagnosis) | Through study completion, an average of 1 per year
  Toronto Extremity Salvage Score (TESS) - Patient functional assessment following for surgery for musculoskeletal tumors (Humeral Reconstruction Stem only) - 100-point score where higher score indicates a better outcome
MSTS (may be used as specific forms related to the pre-operative condition/diagnosis) | Through study completion, an average of 1 per year
  Musculoskeletal Tumor Society (MSTS) - 30 points [6 times (range 0-5)], simple measure of the upper extremity function (Humeral Reconstruction Stem only) - The maximum corresponds to the best score

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Wright, MD, Principal Investigator — UF Health Orthopaedics and Sports Medicine Institute; Young Kwon, MD, Principal Investigator — Hospital for Joint Diseases - NYU Langone Health; Richard Friedman, MD, Principal Investigator — Charleston Orthopaedic Associates; Richard Jones, MD, Principal Investigator — Southeastern Orthopedics and Spine; Howard Routman, DO, Principal Investigator — Florida Atlantis Orthopaedics; Ryan Simovitch, MD, Principal Investigator — Palm Beach Orthopaedic Institute; Geoffrey Abrams, MD, Principal Investigator — Stanford Health Care; Pierre Henri Flurin, MD, Principal Investigator — Centre de l'Arthrose; Yann Marczuk, MD, Principal Investigator — Clinique Chenieux; Harry Brownlow, MD, Principal Investigator — Circle Health Group; Oliver Donaldson, MD, Principal Investigator — Yeovil District Hospital NHS Foundation; Chris Roberts, MD, Principal Investigator — Ipswich Hospital; Chris Peach, MD, Principal Investigator — University Hospital South Manchester; Angelo Di Giunta, MD, Principal Investigator — Policlinico Morgagni; Alfonso Romano, MD, Principal Investigator — Campolongo Hospital; Sean Grey, MD, Principal Investigator — Orthopaedic and Spine Center of the Rockies; Chad Manke, MD, Principal Investigator — Altantic Orthopaedics Specialists; Rick Papandrea, MD, Principal Investigator — Orthopaedic Associates of Wisconsin; Andrew Chambler, MD, Principal Investigator — The Sulis Hospital Bath; Curt Noel, MD, Principal Investigator — Crystal Clinic Orthopaedic; Stephen Parada, MD, Principal Investigator — Orthopedic and Sports Medicine; Ari Youderian, MD, Principal Investigator — South County Orthopedic Specialists; Ian Byram, MD, Principal Investigator — Bone and Joint Institute of Tennessee; Tewfik Benkalfate, MD, Principal Investigator — Clinique Mutualiste la Sagesse; Peter McCann, MD, Principal Investigator — Lenox Health Greenwich Village; Stephanie Muh, MD, Principal Investigator — Henry Ford Health; Bradley Schoch, MD, Principal Investigator — Mayo Clinic; Stephan Pill, MD, Principal Investigator — Steadman Hawkins Clinic of the Carolinas; Scott Trenhaile, MD, Principal Investigator — OrthoIllinois; Bryan Butler, MD, Principal Investigator — Orthopaedic Medical Group of Tampa Bay; Ben Gooding, MD, Principal Investigator — Nottingham City Hospital; Brad Carofino, MD, Principal Investigator — Altantic Orthopaedics Specialist; Ben Sears, MD, Principal Investigator — Western Orthopaedics; Kenneth Faber, MD, Principal Investigator — St Joseph's Health Care; Jaicharan Iyengar, MD, Principal Investigator — Alpine Orthopaedic Medical Group; Oke Anakwenze, MD, Principal Investigator — Duke Department of Orthopedic Surgery; Thomas Obermeyer, MD, Principal Investigator — Barrington Orthopedic; Alison Armstrong, MD, Principal Investigator — Leicester General Hospital; George Malal, MD, Principal Investigator — Bedford Hospital
Locations (38):
- United States (24):
  - South County Orthopedic Specialists, Laguna Woods, California
  - Stanford Health Care, Redwood City, California
  - Alpine Orthopaedic Medical Group, Stockton, California
  - Western Orthopaedics, Denver, Colorado
  - Orthopaedic and Spine Center of the Rockies, Fort Collins, Colorado
  - UF Health Orthopaedics and Sports Medicine Institute, Gainesville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Palm Beach Orthopaedic Institute, Palm Beach Gardens, Florida
  - Florida Atlantis Orthopedics, Palm Beach Gardens, Florida
  - Orthopaedic Medical Group of Tampa Bay, Tampa, Florida
  - Orthopedic and Sports Medicine, Augusta, Georgia
  - OrthoIllinois, Rockford, Illinois
  - Barrington Orthpedic Specialists, Schaumburg, Illinois
  - Henry Ford Health, Detroit, Michigan
  - Hospital for Joint Diseases - NYU Langone Health, New York, New York
  - Lenox Health Greenwich Village, New York, New York
  - Southeastern Sports Medicine and Orthopedics, Asheville, North Carolina
  - Duke Department of Orthopedic Surgery, Durham, North Carolina
  - Crystal Clinic Orthopaedic, Akron, Ohio
  - Charleston Orthopaedic Associates, Charleston, South Carolina
  - Steadman Hawkins Clinic of the Carolinas, Greenville, South Carolina
  - Bone and Joint Institute of Tenessee, Franklin, Tennessee
  - Atlantic Orthopaedics Specialists, Virginia Beach, Virginia
  - Orthopaedic Associates of Wisconsin, Pewaukee, Wisconsin
- St Joseph's Health Care, London, Ontario, Canada
- France (3):
  - Clinique Chenieux, Limoges
  - Centre de l'arthrose, Mérignac
  - Clinique Mutualiste La Sagesse, Rennes
- Italy (2):
  - Policlinico Morgagni, Catania
  - Campolongo Hospital, Eboli
- United Kingdom (8):
  - Circle Health Group, Reading, Berks
  - Yeovil District Hospital NHS Foundation Trust, Yeovil, Summerset
  - The Sulis Hospital Bath, Bath
  - Bedford Hospital, Bedford
  - Ipswich Hospital, Ipswich
  - Leicester General Hospital, Leicester
  - University Hospital South Manchester, Manchester
  - Nottingham University Hospital, Nottingham